CLINICAL TRIAL: NCT02639650
Title: A Prospective Randomized Multicenter Clinical Control Study of Paclitaxel Plus Cisplatin as the First-line Chemotherapy in High Risk Gestational Trophoblastic Tumor
Brief Title: Study of Paclitaxel Plus Cisplatin as the First-line Chemotherapy in High Risk Gestational Trophoblastic Tumor
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Weiguo Lv (Other)
Collaborators: Shandong University (Other); Huazhong University of Science and Technology (Other); First Affiliated Hospital of Zhongshan Medical University (Other)
Responsible Party: Sponsor-Investigator, Weiguo Lv, Vice-President, Women's Hospital School Of Medicine Zhejiang University
Organization: Women's Hospital School Of Medicine Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJHGTN1211
Record Dates: First submitted 2015-12-13; First posted 2015-12-24 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Gestational Trophoblastic Neoplasms
Keywords: gestational trophoblastic tumor; paclitaxel; cisplatin; carboplatin; chemotherapy
MeSH Terms: conditions — Gestational Trophoblastic Disease | interventions — Etoposide; Dactinomycin; Methotrexate; Vincristine; Cyclophosphamide; Paclitaxel; Cisplatin; Carboplatin

ARMS (2):
- control group (Active Comparator): etoposide, methotrexate ,actinomycin D,vincristine, cyclophosphamide(EMA-CO), two weeks a cycle
  Interventions: Drug: Etoposide; Drug: actinomycin D; Drug: methotrexate; Drug: vincristine; Drug: cyclophosphamide
- study group (Experimental): paclitaxel + cisplatin or carboplatin，two weeks a cycle
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Etoposide — etoposide 100mg/m2 ivgtt started at the first day of cycle, two weeks a cycle
  Other Names: VP-16
  Arms: control group
Drug: actinomycin D — actinomycin D 500ug ivgtt, started at the first day of cycle, two weeks a cycle
  Other Names: ACTD; Sanamycin
  Arms: control group
Drug: methotrexate — methotrexate 100mg/m2, 200mg/m2, ivgtt, tetrahydrofolic acid （FA) 15mg q12h*4(24h after methotrexate injection),started at the first day of cycle, two weeks a cycle
  Other Names: MTX
  Arms: control group
Drug: vincristine — vincristine 1mg/m2 started at the 8th day of cycle, two weeks a cycle
  Other Names: VCR
  Arms: control group
Drug: cyclophosphamide — cyclophosphamide 600mg/m2, started at the 8th day of cycle, two weeks a cycle
  Other Names: CTX
  Arms: control group
Drug: Paclitaxel — paclitaxel 135mg/m2, started at the first day of cycle, two weeks a cycle
  Other Names: Taxol
  Arms: study group
Drug: Cisplatin — cisplatin 50mg/m2, started at the first day of cycle, two weeks a cycle
  Other Names: DDP
  Arms: study group
Drug: Carboplatin — carboplatin area under curve (AUC)=4-5, started at the first day of cycle, two weeks a cycle,as a substitute drug for cisplatin
  Other Names: CBP
  Arms: study group

SUMMARY:
This clinical trial is designed to study the effect and safety of paclitaxel plus cisplatin as the first-line regimen in the treatment of high risk gestational trophoblastic tumor.

DETAILED DESCRIPTION:
Gestational trophoblastic tumor (GTN) is a group of malignant tumors derived from placental trophoblastic cells, most of which occur in women of reproductive age. The survival rate of patients with score of 7 or more points, or WHO Ⅳ period for high-risk patients was of 60% to 80%. However, due to severe toxic reactions, long treatment time, loss of optimal reproductive age and increased costs, and treatment failure caused by chemotherapy resistance, high-risk GTN is still one of the tumors seriously affecting the life health and quality of life of young women.

First-line chemotherapy recommended by FIGO is regimen of EMA - CO with corresponding side effects and adverse factors in the following aspects as relatively higer incidence of myelosupression, VP - 16 being associated with a second tumor, especially leukemia, and a definite effect of cyclophosphamide on the failure ovarian function Taxol (Taxol) is the most widely used and most effective broad-spectrum anti-tumor drug in gynecological malignant tumors at present, and T (paclitaxel) +P (platinum drugs) scheme is the first-line chemotherapy scheme in ovarian cancer patients at present. According to references, TP also has effects on resistant and refactory high risk GTN patients.

Given relatively simple operation way of TP chemotherapy, and the effect of chemotherapy in recurrence and high-risk refractory GTN performance,this prospective multicenter randomized controlled clinical research was to study the effect and safety of paclitaxel plus cisplatin as the first-line regimen in the treatment of high risk gestational trophoblastic tumor compared with EMA-CO.

ELIGIBILITY:
Inclusion Criteria:

* Patients who International Federation of Gynecology and Obstetrics (FIGO) Stage I, II, or III criteria for high-risk gestational trophoblastic neoplasia (GTN) and stage Ⅳ cases
* World Health Organization(WHO) risk score ≥7, and less than 13
* Age≤60 years; female, Chinese women
* Initial treatment is chemotherapy
* Performance status: Karnofsky score≥60
* Laboratory tests: WBC≥3.5×10(9)/L, ANC≥1.5×10(9)/L, PLT≥80×10(9)/L, serum bilirubin≤ 1.5 times the upper limit of normal, transaminase≤ 1.5 times the upper limit of normal,blood urea nitrogen, Cr≤ normal
* Provide written informed consent.

Exclusion Criteria:

* Patients with unconfirmed diagnosis of GTN
* Patients with placental-site trophoblastic tumor (PSTT) or epithelioid trophoblastic tumor (ETT)
* WHO risk score less than 7
* With severe or uncontrolled internal disease, unable to receive chemotherapy
* Concurrently participating in other clinical trials
* Unable or unwilling to sign informed consents
* Unable or unwilling to abide by protocol

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 214 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
complete remission rate in firstline treatment | 3 years
  We may calculate the rate of complete response and the rate of treatment failure at the preliminary end point of the trail.

SECONDARY OUTCOMES:
Severity of adverse events as assessed by the WHO | 3 years
  We calculate the adverse events during and after chemotherapy.
Overall Survival Rate (OR) | 3 years
  We calculate the overall survival rate of high risk GTN patients after chemotherapy.
Ovarian functional evaluation | every 6 months up to 3 years
  We may test serum level of anti-mullerian hormone (AMH) every 6 months and the time of menstrual cycle resuming after chemotherapy.
The pregnancy rate | 3 years
  To calculate the pregnancy rate in an actuarial manner using the Kaplan-Meier method at the end of the trail

CONTACTS AND LOCATIONS:
Locations (1):
- Weiguo Lv, Hangzhou, Zhejiang, China